CLINICAL TRIAL: NCT05135221
Title: Combining Biological Therapies in Patients With Inflammatory Bowel Disease: a Finnish Multi-centre Study.
Brief Title: Combination Therapy With Two Biologicals
Acronym: Combi
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Heli T Eronen, Principal investigator, Tampere University Hospital
Other Study IDs: CBT
Record Dates: First submitted 2021-10-13; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: IBD
Keywords: biological; combination therapy; adalimumab; ustekinumab; vedolizumab; golimumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: dual biological therapy — Simultaneous use of two biologicals.

SUMMARY:
The efficacy and safety of dual biological therapy.

DETAILED DESCRIPTION:
Data of all patients treated with the combination of two biologicals in four Finnish tertiary centres were collected and analysed. Inclusion criteria were simultaneous use of two biological treatments (infliximab, adalimumab, golimumab, vedolizumab or ustekinumab), age 16 years or over and follow-up for at least induction period after introduction of second biological therapy. The primary outcome was effectiveness, defined as remission assessed by physician after at least four months of DBT. The secondary outcome was safety defined by any adverse events or infection complications during DBT.

ELIGIBILITY:
Inclusion Criteria:

* Simultaneous use of two different biological treatments for IBD.
* Treatment duration with combination therapy for at least for induction period.

Exclusion Criteria:

-Age under 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients treated in Finnish tertiary centers.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical response | 18 months
  In CD, clinical response was assessed using a modified Harvey-Bradshaw index (HBI, omitting abdominal palpation) and clinical remission was defined as HBI<5. In UC, partial MAYO score <3 was cut the off value for clinical remission. Patients symptoms were assessed at baseline, 4, 12 and 18 months after initiation of treatment.

SECONDARY OUTCOMES:
Endoscopic response | 18 months
  Endoscopic response was assessed by Mayo endoscopic score for UC, simple endoscopic score for CD based on endoscopic characteristics (MAYO ≤ 1 and SES-CD < 3 as cut off values for endoscopic remission). Endoscopy was performed at baseline and 4, 12 or 18 months after initiation of treatment.
Haemoglobin level improvement | 18 months
  Blood haemoglobin ≥117 g/L for females and ≥134 g/L for males. Measured at baseline and 4, 12 and 18 months after initiation of treatment.
Calprotectin level improvement | 18 months
  Change in fecal Calprotectin level measured from baseline and 4, 12 and 18 months of treatment. Feacal calprotectin level ≤ 250 µg/g as cut-off value for remission.
C-reactive protein level improvement. | 18 months
  CRP < 10 mg/L. CRP levels were measured at baseline and 4, 12 and 18 months after initiation of treatment.
Treatment related infections | 18 months
  Infection complications reported during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Heli Eronen, Principal Investigator — Kanta-Häme Central Hospital
Locations (1):
- Heli Eronen, Lempäälä, Finland

IPD SHARING:
Plan to Share IPD: No